CLINICAL TRIAL: NCT01225445
Title: Treatment of Early Immunoglobulin A Nephropathy by Angiotensin Converting Enzyme Inhibitor - A Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Cheuk Chun Szeto, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE 498/6015
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2002-04

CONDITIONS: Biopsy-confirmed IgA Nephropathy; Proteinuria Less Than 0.5 g Per Day; Normal Blood Pressure; Serum Creatinine Below 120 Umol/l
MeSH Terms: interventions — Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): ramipril 2.5 mg daily
  Interventions: Drug: Ramipril
- Control (No Intervention)

INTERVENTIONS:
Drug: Ramipril — 2.5 mg daily
  Arms: Treatment

SUMMARY:
Immunoglobulin A (IgA) nephropathy is the most common type of primary glomerulonephritis in the world. The treatment of IgA nephropathy with normal renal function and minimal proteinuria is unknown. Since angiotensin-converting enzyme (ACE) inhibitors reduce proteinuria and retard the rate of decline of renal function in chronic proteinuric nephropathies, including IgA nephropathy. The investigators conduct a randomized control study to evaluate the efficacy of ACE inhibitor in the treatment of early IgA nephropathy. Sixty patients with biopsy-proven IgA nephropathy and minimal proteinuria are recruited. They will be randomized to ramipril for 5 years or no treatment. Blood pressure, proteinuria and renal function will be monitored. This study will explore the effects of ACE inhibitor in the treatment of early IgA nephropathy, which is a major cause of dialysis-dependent renal failure.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65
* biopsy-confirmed IgA nephropathy
* proteinuria less than 0.5 g per day, normal blood pressure, and serum creatinine below 120 umol/l
* willingness to give written informed consent and willingness to participate in and comply with the study protocol

Exclusion Criteria:

* expected survival less than 2 years
* pregnant or nursing mother, or women of childbearing potential without an effective method of birth control
* history of myocardial infarction, congestive heart failure, or any other medical indication that necessitate the use of ACE inhibitor
* evidence of clinically significant hepatic, gastrointestinal, autoimmune disease
* history of malignancy, drug or alcohol abuse
* participation in any previous trial on ACE inhibitor
* taking other investigational drugs within the past 30 days
* history of non-compliance to medical regimens and patients who are considered potentially unreliable
* known history of sensitivity / allergy to ACE inhibitor

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2002-04; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
blood pressure | 5 years
proteinuria | 5 years
  over 1 g/day
serum creatinine | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Cheuk Chun Szeto, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Medicine & Therapeutics, Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639